CLINICAL TRIAL: NCT00569920
Title: Nausea and Pain Prophylaxis During Thyroid Surgery, a Comparison of Low-Dose and High-Dose Dexamethasone to Placebo
Brief Title: Nausea and Pain Prophylaxis During Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Telemark (Other Government)
Responsible Party: Simen Doksrød/Acting chief physician, Sykehuset Telemark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: s8197.04; S-04189
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: Thyroid Diseases; Parathyroid Diseases
MeSH Terms: conditions — Thyroid Diseases; Parathyroid Diseases | interventions — Dexamethasone; dexamethasone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: natriumchloride 0,9%
- 2 (Active Comparator): dexamethasone "low-dose"
  Interventions: Drug: dexamethasone
- 3 (Active Comparator): Dexamethasone "high-dose"
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: dexamethasone — IV dexamethasone 0,15 mg/kg bodyweight. Single-dose bolus injection after start of anesthesia. Medication is opened and administrated to the patient from a coded ampoule by the physician. The medication is diluted in such a way that 1 mL is equivalent to 10 kg body weight (1,5 mg/mL).
  Other Names: Fortecortin
  Arms: 2
Drug: natriumchloride 0,9% — iv natriumchloride 0,9% (placebo). 1 mL is equivalent to 10 kg body weight.
  Arms: 1
Drug: dexamethasone — IV dexamethasone 0,30 mg/kg body weight. Drug diluted to 3,0 mg/mL and administrated in same way as arm 2.
  Other Names: fortecortin
  Arms: 3

SUMMARY:
Postoperative pain and nausea may diminish a patient's wellbeing, and may also delay rehabilitation, as well as increase the total cost of care and treatment. Opioids are effective drugs for treatment of pain, but with the disadvantage of side effects such as somnolence and nausea. The benefits of various types of non-opioid analgesic in reducing patients' postoperative need for opioids have been well-documented.

One non-opioid prophylaxis documented for various surgery is short-term treatment with corticosteroids. The optimal dose of corticosteroids for peroperative nausea and pain prophylaxis is not well-documented. In our study we will attempt to determine whether the aforementioned benefits of corticosteroids are valid for a group of patients undergoing thyroid surgery.

Hypothesis: Single-dose treatment with dexamethasone provides a better analgesic effect and/or reduced use of opioids than placebo in patients undergoing elective throid surgery. Higher dose of dexamethasone provide better and/or longer-lasting analgesic effects without influencing the side effect profile.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients scheduled for elective thyroid surgery and parathyroid surgery under general anesthesia.
* Informed consent

Exclusion Criteria:

* Patients who use steroids
* Patients who use antiemetics
* Patients who use opioid analgesics
* Body weight > 100 kg
* BMI > 35

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pain (VAS) and use of opioids. Nausea. | 30 days

SECONDARY OUTCOMES:
Nausea | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Johan Raeder, Prof. M.D, Study Director — Ullevål university hospital, Oslo university
Locations (1):
- Surgery Unit, Porsgrunn, Acute Care Clinic, Telemark Hospital, Porsgrunn, Telemark, Norway